CLINICAL TRIAL: NCT05638282
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Subcutaneous Doses of Cendakimab in Chinese Healthy Participants
Brief Title: A Study to Evaluate the Safety and Tolerability of Cendakimab in Chinese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM042-005
Record Dates: First submitted 2022-11-30; First posted 2022-12-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy Participants
Keywords: Healthy; Chinese; Cendakimab
MeSH Terms: interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cendakimab (Experimental)
  Interventions: Drug: Cendakimab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cendakimab — Specified dose on specified days
  Other Names: CC-93538, BMS-986355, RPC4046
  Arms: Cendakimab
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the drug levels, safety, and tolerability of cendakimab in healthy male and female Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Chinese (both biological parents are ethnically Chinese).
* Body mass index (BMI) of 18.0 through 28.0 kilograms/meter squared (kg/m^2), inclusive. BMI = weight (kg)/[height (m)]^2.
* Body weight ≥ 50.0 kg.

Exclusion Criteria:

* History of clinically significant infection within 4 weeks of dosing on Day 1.
* Significant medical history/condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
* Condition(s) which may confound the ability to interpret data from the study, as determined by the investigator.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Predose and at multiple timepoints (up to 105 days) after dosing
Area Under the Serum Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) | Predose and at multiple timepoints (up to 105 days) after dosing
Area Under the Serum Concentration-time Curve from Time Zero Extrapolated to Infinite Time (AUC(INF)) | Predose and at multiple timepoints (up to 105 days) after dosing

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Day 1 through Day 105
Number of Participants with Clinically Significant Changes in Clinical Laboratory Tests | Screening (Days -28 to -1) through Day 105
Number of Participants with Clinically Significant Changes in Vital Signs | Screening (Days -28 to -1) through Day 105
Number of Participants with Clinically Significant Changes in Physical Examinations | Screening (Days -28 to -1) through Day 105
Number of Participants with Clinically Significant Changes in Electrocardiograms | Screening (Days -28 to -1) through Day 105

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com